CLINICAL TRIAL: NCT01879969
Title: Computer Assisted Orthognathic Surgery. Facial Asymmetry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Responsible Party: Principal Investigator, Silvio Mario Meloni, DDS, PhD, Assistant Professor, Università degli Studi di Sassari
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDM 06/06/13
Record Dates: First submitted 2013-06-06; First posted 2013-06-18 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Facial Asymmetry
Keywords: computer-assisted orthognathic surgery; facial asymmetry
MeSH Terms: conditions — Facial Asymmetry

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- asymmetric patients, classic procedure (Experimental): random selected
  Interventions: Procedure: classic procedure of planning
- asymmetric patients, computer assisted (Experimental): random selected
  Interventions: Procedure: computer assisted orthognathic planning and surgery of asymmetric patients

INTERVENTIONS:
Procedure: classic procedure of planning — analysis of pictures, 2D radiographs and aesthetics; model surgery and acrylic splint
  Arms: asymmetric patients, classic procedure
Procedure: computer assisted orthognathic planning and surgery of asymmetric patients
  Other Names: CBCT, data acquisition and processing; virtual surgery and CAD/CAM intermediate splint
  Arms: asymmetric patients, computer assisted

SUMMARY:
The specific aims of the study were to measure and compare the rates of alignment and cant reduction of the dental and facial midlines among the two groups.

DETAILED DESCRIPTION:
The purpose of this randomized, controlled, clinical study, was to evaluate the most accurate procedure for orthognathic correction of facial asymmetry. The investigators compared two different methods of surgical planning: classical (esthetic analysis of the face, cephalometric study of the skull in lateral and posteroanterior cephalograms, analysis and surgical simulation of plaster casts mounted in semi-individual articulators, development of a surgical acrylic resin intermediate splint) and digital planning (cone-beam computed tomography, data acquisition, software-assisted virtual surgery -Maxilim; Medicim, Mechelen, Belgium- and CAD/CAM processing of the surgical intermediate splint).

ELIGIBILITY:
Inclusion Criteria:

* facial asymmetry or mandibular deviation (cant of the occlusal plane > 3° and/or midline discrepancies > 2.5 mm)
* presence of all central incisors,
* pre- and postoperative radiographs and plaster casts (group 1)
* cranial CBCT images (group 2)
* pre- and postoperative digital photographs.

Exclusion Criteria:

* previous trauma involving the hard or soft facial tissues
* functional deviation of the mandible
* incomplete records (CBCT, radiographs, casts or digital photographs).

Ages: 21 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-12; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in linear measures | Preoperative (baseline)-Postoperative (up to 1 month)
  More specifically were measured: distance from the upper interincisal point to the facial midline; distance from the lower interincisal point to the facial midline; distance between interincisal points; distance from skeletal menton to the facial midline; distance from soft tissue menton to the facial midline;
Change in angular measures | Preoperative (baseline)- Postoperative (up to one month)
  More specifically were measured:distance from the maxillary sagittal plane to the facial mid-sagittal plane; distance from the mandibular sagittal plane to the facial mid-sagittal plane.

SECONDARY OUTCOMES:
age of patients | Preoperative (baseline)
  age at surgery
Type of surgery needed | Preoperative (baseline)
  How many patients had genioplasty added to the standard bimaxillary surgery plan
sample size | Preoperative (baseline)
  number of patients
gender | Preoperative (baseline)
  male/female

CONTACTS AND LOCATIONS:
Locations (1):
- Maxillofacial Unit, University of Sassari, Sassari, SS, Italy